CLINICAL TRIAL: NCT02271659
Title: Medical and Economic Evaluation of an External Beam Radiotherapy Combined With a Brachytherapy Boost Compared With an Exclusive External Beam Radiotherapy for Intermediate-risk Prostate Cancer
Brief Title: Medical and Economic Evaluation for Intermediate-risk Prostate Cancer
Acronym: GETUGP05
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-704
Record Dates: First submitted 2014-06-02; First posted 2014-10-22 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Prostate Cancer
Keywords: Prostate; external beam radiotherapy; brachytherapy boost; economical evaluation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brachytherapy boost (Experimental): Brachytherapy boost with external beam radiotherapy. External beam radiotherapy of 46 Gy delivered to the prostate and the first centimeter of the seminal vesicles with a brachytherapy boost (of iodine-125 seeds (110Gy) or high dose rate (14Gy) with iridium-192) only to the prostate. Each center will choose the appropriate brachytherapy technique
  Interventions: Radiation: Brachytherapy boost with external beam radiotherapy
- Exclusive external beam irradiation (Active Comparator): Exclusive external beam radiotherapy. External beam radiotherapy of 46 Gy delivered to the prostate and the first centimeter of the seminal vesicles with an external beam radiotherapy of 80 Gy to the prostate alone.
  Interventions: Radiation: Exclusive external beam radiotherapy

INTERVENTIONS:
Radiation: Brachytherapy boost with external beam radiotherapy — Bras A: External beam radiotherapy of 46 Gy delivered with a linear accelerator (Varian) to the prostate and the first centimeter of the seminal vesicles with a brachytherapy boost (of iodine-125 seeds from Bard (110Gy) or high dose rate (14Gy) with a iridium-192 source) only to the prostate. Each center will choose the appropriate brachytherapy technique. The number of seeds or needles will depend on the prostate's volume.
  Arms: Brachytherapy boost
Radiation: Exclusive external beam radiotherapy — Bras B: External beam radiotherapy of 46 Gy delivered with photons and a linear accelerator (Varian) to the prostate and the first centimeter of the seminal vesicles with an external beam radiotherapy of 80 Gy to the prostate alone.
  Arms: Exclusive external beam irradiation

SUMMARY:
The aim of the present phase III study is two-folded: 1) to show a superiority of external beam radiotherapy combined with a brachytherapy boost versus exclusive external beam radiotherapy and 2) to evaluate the economic impact of each treatment.

The study includes 33 cancer centres, the inclusion time is of 2 years and the follow-up is of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years;
* life expectancy of greater than 10 years;
* prostate adenocarcinoma histologically proven;
* prostate cancer has to be of intermediate-risk based on at least one of the three following criteria: PSA between 10 ng/ml and 20 ng/ml, and/or a Gleason score of 7 and/or a T2B. Karnofsky performance status ≥ 60% and consequently performance status ECOG 0-2.
* the patient has to be the beneficiary of the social security system (order n° 2006-477 from April 26th 2006);
* the signed consent form.

Exclusion Criteria:

* PSA level > 20;
* Gleason > 7;
* clinical T3A or T3B or MRI (a simple suspicion/ doubt on the MRI regarding the T3A won't be an exclusion criterion);
* prostate volume > 60 cc;
* pelvic lymph nodes involvement at dissection or imaging (ADP > 1.5 cm);
* concurrent hormone therapy;
* the presence of distant metastasis (M1);
* history of abdominal or pelvic irradiation;
* history of prostate resection in the previous 6 months and/or not allowing the implantation of markers;
* history of uncontrolled cancer and/or treated since less than 5 years (excepting the basal-cell carcinoma);
* urinary discomfort with an IPSS (International Prostate Symptom Score) > 15 (without alpha-blocking);
* inflammatory bowel disorder such as ulcerative colitis or the Crohn's disease;
* other undergoing study that may interfere with the present study;
* patient under legal protection measure.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2013-06; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the biochemical relapse free survival of the patients in two groups at 5 years for an external beam radiotherapy with a brachytherapy boost versus an exclusive external beam radiotherapy | 5 years
  Biochemical relapse is defined using the Phoenix definition of nadir of Prostate Specific Antigen + 2 ng/ml. This will be studied for both arms

SECONDARY OUTCOMES:
The evaluation of the overall survival at 5 years. | 5 years
  All cause mortality
The evaluation of the specific survival at 5 years | 5 years
  Mortality due to prostate cancer
The evaluation of the survival without any metastatic evolution at 5 years | 5 years
The study of all toxicities | 5 years
  The toxicities include: acute and late toxicities, sexual toxicities, the quality of life of the patients (CTCAE version 4.0)
Medical and economical evaluation. | 5 years
  The complete medical and economical evaluation of the strategies

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHAPET, MD, Principal Investigator — HCL
Locations (29):
- France (29):
  - Clinique Claude Bernard, Albi
  - CHU Jean MINJOZ, Besançon
  - Clinique Tivoli, Bordeaux
  - Institut Bergonie, Bordeaux
  - CHRU Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Hopital de la Tronche, Grenoble
  - Centre Regional de Lutte Contre Le Cancer Rhone-Alpes Centre Leon Berard, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre d'oncologie et de radiothérapie Mâcon, Mâcon
  - Centre Val D'Aurelle, Montpellier
  - Institut de Cancerologie de Lorraine Alexis Vautrin, Nancy
  - Clinique Hartmann, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hopital Saint-Louis, Paris
  - Hopital George Pompidou, Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Institut Jean Godinot,, Reims
  - Polyclinique Courlancy, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henry Becquerel, Rouen
  - Institut Cancérologique de la Loire, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
  - Clinique du TONKIN, Villeurbanne